CLINICAL TRIAL: NCT01551420
Title: Home Study of an Advanced Upper Limb Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0771-R; A9226-R (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2012-02-27; First posted 2012-03-12 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Amputation of Arm
Keywords: Amputation; Prosthetic Design; Upper Extremity

STUDY DESIGN:
Intervention Model Description: Sequential testing in non-equivalent comparison groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Advanced upper limb prosthetic device IMU controlled (Active Comparator): Subjects with upper limb amputation who are trained to use a DEKA Arm with IMU controls
  Interventions: Device: Advanced upper limb prosthetic device IMU controlled
- Advanced upper limb prosthetic EMG-PR controlled (Active Comparator): Subjects with TR or TH upper limb amputation who are trained to use a DEKA Arm with EMG-PR Controls
  Interventions: Device: Advanced upper limb prosthetic EMG-PR controlled

INTERVENTIONS:
Device: Advanced upper limb prosthetic device IMU controlled — Advanced upper limb prosthetic IMU controlled
  Other Names: DEKA Arm, DARPA Arm IMU controlled
  Arms: Advanced upper limb prosthetic device IMU controlled
Device: Advanced upper limb prosthetic EMG-PR controlled — Advanced upper limb prosthetic EMG-PR controlled
  Other Names: DEKA Arm, DARPA Arm EMG-PR controlled
  Arms: Advanced upper limb prosthetic EMG-PR controlled

SUMMARY:
The overall study objective is to examine the feasibility, acceptance, and benefits of home use of an advanced upper limb prosthetic device as well as the logistical support requirements utilized during 3 months of home usage. All participating subjects will enroll in Part A of the study which will involve supervised training. Eligible subjects will be invited to participate in Part B, the home use portion of the study.

DETAILED DESCRIPTION:
The specific objectives of this study are to:

1. identify and describe upper limb amputees who would be appropriate candidates for home use of this advanced prosthesis as well as those who would not be appropriate.
2. Compare the extent of use of the existing prosthesis to that of the DEKA Arm.and quantify the impact of home use of the DEKA Arm on device satisfaction, performance of functional activities and the user's quality of life.
3. Compare the outcomes of users of pattern recognition to the outcomes of users without
4. quantify the amount and type of technical support and repairs needed during the study, and estimate the number of home study days lost due to service/repair.

All participating subjects will enroll in Part A of the study, which will involve supervised, in-laboratory training, as well as supervised community based outings. Based upon the findings from Part A, study staff will classify participants as appropriate or not appropriate for participation in Part B (the home usage portion of the study). Final determination of appropriateness for home use will be made after a home visit. The home use portion of the study will last for 13 weeks and involve regularly scheduled study visits.

Measures of existing prosthetic activity will be compared with those of home use of the advanced upper limb prosthetic device to determine the extent of adoption. Changes in device satisfaction, performance of functional activities, and quality of life will be evaluated throughout the study. Data on technical support usage will also be gathered.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Parts A and B):

* All subjects must be at least 18 years old and have single or bilateral upper limb amputation.
* Subjects must be able to understand the requirements of the study and sign an Informed Consent Form and HIPAA Authorization Form.
* Subjects will include those who are current users of any type of prosthetic device (body powered, electric or hybrid), non-users of devices who have been previously fit with a device, but have chosen not to wear it, as well as new users of devices.
* To participate in the study all subjects must have active control over one or both ankles, OR have an appropriate number of myoelectric and/or other control sites (as determined by the Principal Investigator in conjunction with the research team) to allow adequate prosthetic controls configuration.

Inclusion Criteria Part B only:

* Completion of all Part A study activities.
* Meets all criteria for Preliminary Determination of Appropriateness for Unsupervised, Home Device Use.

Exclusion Criteria:

Exclusion Criteria (Parts A and B):

* Amputees with elbow disarticulation, wrist disarticulation and partial hand amputations will be excluded. *beginning July 1, 2016 amputees with shoulder disarticulation or forequarter amputation will be excluded.
* Amputees will be excluded if the length of their residual limb would prohibit socket fitting, as determined by the study prosthetist.
* Persons with significant uncorrectable visual deficits that would impair the ability to see the prosthesis and those who have major communication or neurocognitive deficits will be excluded.
* Persons with skin conditions such as burns or poor skin coverage as well as those with severe contractures that prevented prior prosthetic wear will be excluded.
* Persons with electrically controlled medical devices including pacemakers, and implanted defibrillators will be excluded.
* Persons with neuropathy, uncontrolled diabetes, who are receiving dialysis, have insensate feet, severe phantom pain or a history of skin ulcers or any other significant comorbidity which would interfere with the study will be excluded.
* Those with severe circulatory problems including peripheral vascular disease and pitting edema will be excluded.
* Persons with cognitive deficits or mental health problems that would limit their ability to participate fully in the study protocol will be excluded.
* Women who are pregnant or who plan to become pregnant in the near future will also be excluded.
* The investigators will exclude those amputees who work for prosthetic companies that may be considered competitors for the prosthetic arm technology in the future.
* Persons taking medication which poses a risk for operation of heavy equipment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Center for the Intrepid/ Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resnik L, Borgia M, Acluche F. Brief activity performance measure for upper limb amputees: BAM-ULA. Prosthet Orthot Int. 2018 Feb;42(1):75-83. doi: 10.1177/0309364616684196. Epub 2017 Jan 16. PMID 28091278
- [Background] Resnik L, Borgia M, Acluche F. Timed activity performance in persons with upper limb amputation: A preliminary study. J Hand Ther. 2017 Oct-Dec;30(4):468-476. doi: 10.1016/j.jht.2017.03.008. Epub 2017 May 6. PMID 28487130
- [Background] Resnik LJ, Borgia ML, Acluche F. Perceptions of satisfaction, usability and desirability of the DEKA Arm before and after a trial of home use. PLoS One. 2017 Jun 2;12(6):e0178640. doi: 10.1371/journal.pone.0178640. eCollection 2017. PMID 28575025
- [Background] Resnik L, Fantini C, Latlief G, Phillips S, Sasson N, Sepulveda E. Use of the DEKA Arm for amputees with brachial plexus injury: A case series. PLoS One. 2017 Jun 19;12(6):e0178642. doi: 10.1371/journal.pone.0178642. eCollection 2017. PMID 28628623
- [Background] Resnik L, Acluche F, Borgia M. The DEKA hand: A multifunction prosthetic terminal device-patterns of grip usage at home. Prosthet Orthot Int. 2018 Aug;42(4):446-454. doi: 10.1177/0309364617728117. Epub 2017 Sep 15. PMID 28914583
- [Background] Resnik L, Acluche F, Lieberman Klinger S, Borgia M. Does the DEKA Arm substitute for or supplement conventional prostheses. Prosthet Orthot Int. 2018 Oct;42(5):534-543. doi: 10.1177/0309364617729924. Epub 2017 Sep 14. PMID 28905665
- [Background] Resnik L, Klinger S. Attrition and retention in upper limb prosthetics research: experience of the VA home study of the DEKA arm. Disabil Rehabil Assist Technol. 2017 Nov;12(8):816-821. doi: 10.1080/17483107.2016.1269212. Epub 2017 Jan 18. PMID 28098513
- [Background] Resnik, L. Cancio, J. Fantini, C. Ikeda, A. Sasson, N. Pattern Recognition Control of the DEKA Arm in Two Transhumeral Amputees with Target Muscle Reinnervation, Conference Proceedings, Myoelectric Control Conference (MEC), 2017
- [Result] Resnik L, Cancio J, Klinger S, Latlief G, Sasson N, Smurr-Walters L. Predictors of retention and attrition in a study of an advanced upper limb prosthesis: implications for adoption of the DEKA Arm. Disabil Rehabil Assist Technol. 2018 Feb;13(2):206-210. doi: 10.1080/17483107.2017.1304585. Epub 2017 Apr 4. PMID 28375687
- [Result] Resnik LJ, Borgia ML, Acluche F, Cancio JM, Latlief G, Sasson N. How do the outcomes of the DEKA Arm compare to conventional prostheses? PLoS One. 2018 Jan 17;13(1):e0191326. doi: 10.1371/journal.pone.0191326. eCollection 2018. PMID 29342217
- [Result] Resnik L, Klinger S, Gill A, Ekerholm Biester S. Feminine identity and functional benefits are key factors in women's decision making about upper limb prostheses: a case series. Disabil Rehabil Assist Technol. 2019 Feb;14(2):194-208. doi: 10.1080/17483107.2018.1467973. Epub 2018 May 9. PMID 29741966
- [Result] Resnik L, Acluche F, Borgia M, Cancio J, Latlief G, Sasson N. Function, quality of life, and community integration of DEKA Arm users after discharge from prosthetic training: Impact of home use experience. Prosthet Orthot Int. 2018 Dec;42(6):571-582. doi: 10.1177/0309364618774054. Epub 2018 May 19. PMID 29779455
- [Result] Resnik LJ, Acluche F, Lieberman Klinger S. User experience of controlling the DEKA Arm with EMG pattern recognition. PLoS One. 2018 Sep 21;13(9):e0203987. doi: 10.1371/journal.pone.0203987. eCollection 2018. PMID 30240420
- [Result] Resnik LJ, Acluche F, Borgia M, Cancio J, Latlief G, Phillips S, Sasson N. EMG pattern recognition compared to foot control of the DEKA Arm. PLoS One. 2018 Oct 18;13(10):e0204854. doi: 10.1371/journal.pone.0204854. eCollection 2018. PMID 30335781

RESULTS

PARTICIPANT FLOW:
Period: In-laboratory (Part A)
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Started | 39 | 13
Completed | 33 | 11
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Scheduling conflict | 2 | 1
Period: Screened for Part B Eligibility
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Started | 33 | 11
Completed | 24 | 8
Not Completed | 9 | 3
Not completed — Declined participation | 8 | 1
Not completed — Deemed ineligible by staff | 1 | 2
Period: Home Use (Part B)
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Started | 24 | 8
Completed | 18 | 7
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Withdrawal by staff | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled | Total
Number analyzed (Participants) | 39 | 13 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 11 | 43
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (16.1) | 46.1 (15.4) | 45.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 34 | 11 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 32 | 12 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 31 | 13 | 44
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life (QOL) Scale
Description: The QOL consists of 16 questions that assess satisfaction with independent living and self-care activities. Each item is rated (1=Terrible to 7=Delighted). The average of these 16 items is the summary score with higher values reflecting higher satisfaction. The primary outcome is the net change in summary score between baseline and end of Part B.
Time Frame: baseline and after 9-12 weeks of home use (end of Part B)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 17 | 7
score on a scale | 5.8 (0.7) | 5.3 (0.6)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Test type: Superiority — Null hypothesis of no change after home use; p = .9358, t-test, 2 sided — Two way comparison between scores at baseline and after 9-12 weeks of Prosthetic use. Alpha=0.05; paired t-tests; Mean Difference (Net) = .002, 95% CI 2-sided [-0.27 to 0.28], Standard Deviation 0.68
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of QOL measure at 9-12 weeks, comparing groups by control type, controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.08, Regression, Linear; Slope = -0.69, 95% CI 2-sided [-1.47 to 0.09]

2. Secondary Outcome: Upper Extremity Functional Scale (UEFS) From the Orthotics and Prosthetics Users Survey (OPUS) Use Scale
Description: Measures the engagement of the prosthesis in everyday activities using 23 items from the OPUS UEFS. Respondents indicate which activities they performed using a prosthesis. The score is the proportion of activities performed using a prosthesis.
Time Frame: Baseline, end of Part A (variable time frame depending on training schedule), after 9-12 weeks of home use (end of Part B)
Population: Prosthesis users only, at baseline, completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: proportion of activities performed
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 39 | 13
proportion of activities performed
  Prosthesis users at baseline | 0.3 (0.3) | 0.4 (0.3)
  Completers End of Part A: number analyzed (Participants) | 33 | 11
  Completers End of Part A | 0.7 (0.3) | 0.6 (0.3)
  Completers End of B: number analyzed (Participants) | 18 | 7
  Completers End of B | 0.6 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e participants with UEFS data at both time points); Test type: Superiority; p < 0.0001, t-test, 2 sided; The sample for this analyses was 44 participants; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.17 to 0.43], Standard Deviation 0.42 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from UEFS use measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p < 0.0001, Regression, Linear; The sample for this analysis was 23 participants with TR or TH amputation level who completed data collection for UEFS at End of Part B; Slope = -0.56, 95% CI 2-sided [-0.73 to -0.40], Standard Error of Mean 0.08 — Effect of EMG-PR (compared to IMU group)

3. Secondary Outcome: Trinity Amputations and Prosthetics Experience Scale (TAPES) Satisfaction Scale
Description: The TAPES Satisfaction scale is a 10-item scale measuring extent of satisfaction regarding functional characteristics of the artificial limb: reliability, comfort, fit, and overall satisfaction, contentment with cosmetic characteristics of the device. Each item is rated from 1-5 (1=Very Dissatisfied to 5=Very Satisfied). The average score is used.
Time Frame: as for outcome 2
Population: Prosthesis users only, at baseline, completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 33 | 12
score on a scale
  Prosthesis users at baseline: number analyzed (Participants) | 28 | 12
  Prosthesis users at baseline | 3.6 (0.7) | 3.7 (0.8)
  Completers End of Part A: number analyzed (Participants) | 33 | 11
  Completers End of Part A | 3.5 (0.7) | 3.0 (0.6)
  Completers End of B: number analyzed (Participants) | 18 | 7
  Completers End of B | 3.8 (0.9) | 2.7 (1.1)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e participants with TAPES data at both time points); Test type: Superiority; p = 0.186, t-test, 2 sided; The sample for this analysis was 34 participants; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.55 to 0.11], Standard Deviation 0.94 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from TAPES measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0168, Regression, Linear; The sample for this analysis was 24 participants with TR or TH amputation level who completed data collection for TAPES at End of Part B; Slope = -1.15, 95% CI 2-sided [-2.06 to -0.23], Standard Error of Mean 0.44 — Effect of EMG-PR (compared to IMU group)

4. Secondary Outcome: Activities Measure for Upper Limb Amputees (AM-ULA)
Description: The AM-ULA is an 18-item measure assessing functional performance with a prosthesis: ability of the amputee to complete daily activities, speed of the performance, movement quality, skillfulness of prosthetic use and independence. Items are rated 0=Unable to perform task to 4=Excellent Performance. Average score is multiplied by 10 and has a range from 0 (lowest functional performance) to 40 (highest functional performance).
Time Frame: as for outcome 2
Population: Prosthesis users only, at baseline, completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 33 | 11
units on a scale
  Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  Prosthesis users at baseline | 17.5 (6.1) | 10.4 (3.3)
  Completers End of Part A | 16.8 (4.5) | 16.8 (3.1)
  Completers End of B: number analyzed (Participants) | 16 | 7
  Completers End of B | 10.7 (4.4) | 19.8 (1.8)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with UEFS data at both time points); Test type: Superiority; p = 0.3367, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -0.97, 95% CI 2-sided [-2.99 to 1.05], Standard Deviation 5.61 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from AM-ULA measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.6339, Regression, Linear; The sample for this analysis was 22 participants with TR or TH amputation level who completed data collection for UEFS at End of Part B; Slope = -0.72, 95% CI 2-sided [-3.84 to 2.39], Standard Error of Mean 1.49 — Effect of EMG-PR (compared to IMU group)

5. Secondary Outcome: Three Scales of the Veterans Version of the SF-36
Description: Role Physical: measures role physical function with 4 items referring to role limitations due to physical health. Items are rated from 1=none of the time to 5=All of the time. Social Functioning: measures social functioning with 2 items referring to problems interfering with socializing with friends and family. One item is rated extent of problems as 1=Not at all to 5=Extremely and is reverse coded. All other items are rated as problem frequency from 1=All of the time to 5=None of the time. The mean score is scaled to range between 0 to 100. Physical Functioning: measures physical functioning with 10 items pertaining to moving, lifting and walking. Items are rated from 1=Limited a lot to 3=Not limited at all. The mean score is scaled to range between 0 to 100. In all scales, higher scores correspond to higher quality of life.
Time Frame: as for outcome 2
Population: Baseline participants and completers at End of A and End of B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 39 | 13
score on a scale
  Role Physical: Participants at Baseline | 80.0 (18.8) | 74.5 (24.3)
  Role Physical:Completers at End of Part A: number analyzed (Participants) | 33 | 10
  Role Physical:Completers at End of Part A | 77.8 (21.5) | 71.3 (25.7)
  Role Physical: Completers at End of B: number analyzed (Participants) | 19 | 7
  Role Physical: Completers at End of B | 82.2 (17.7) | 72.3 (22.2)
  Social Functioning: Participants at Baseline | 88.5 (18.0) | 86.5 (13.9)
  Social Functioning: Completers at End of Part A: number analyzed (Participants) | 33 | 10
  Social Functioning: Completers at End of Part A | 86.4 (23.3) | 77.5 (19.4)
  Social Functioning: Completers End of B: number analyzed (Participants) | 19 | 7
  Social Functioning: Completers End of B | 86.8 (15.9) | 80.4 (18.9)
  Physical Functioning: Participants at Baseline | 82.6 (15.8) | 68.8 (22.5)
  Physical Functioning: Completers at End of Part A: number analyzed (Participants) | 33 | 10
  Physical Functioning: Completers at End of Part A | 80.4 (18.2) | 68.5 (24.2)
  Physical Functioning: Completers at End of B: number analyzed (Participants) | 19 | 7
  Physical Functioning: Completers at End of B | 82.6 (18.4) | 55.7 (15.4)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data for participants at baseline and completers at End of A (i.e participants with SF-36V Role Physical data at both time points); Test type: Superiority; p = 0.5465, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -1.74, 95% CI 2-sided [-7.53 to 4.05], Standard Deviation 18.8 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data for participants at baseline to End of A (with SF-36V Social Functioning data at both time points); Test type: Superiority; p = 0.1610, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -3.78, 95% CI 2-sided [-9.12 to 1.57], Standard Deviation 17.37 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 3: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data for participants at baseline to End of A (with SF-36V Physical Functioning data at both time points); Test type: Superiority; p = 0.7765, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -0.61, 95% CI 2-sided [-4.90 to 3.68], Standard Deviation 13.9 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 4: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of SF-36V; Role Physical measure at 9-12 weeks, comparing groups by control type, controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0669, Regression, Linear; The sample for this analysis was 23 participants with TR or TH amputation level who completed data collection for SF-36 at End of Part B; Slope = -13.35, 95% CI 2-sided [-27.72 to 1.02], Standard Error of Mean 6.91 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 5: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of SF-36V: Social Functioning measure at 9-12 weeks, comparing groups by control type, controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.2592, Regression, Linear; [statistical method as in outcome 5, analysis 4]; Slope = -8.24, 95% CI 2-sided [-23.01 to 6.54], Standard Error of Mean 7.10 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 6: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of SF-36V: Physical Functioning measure at 9-12 weeks, comparing groups by control type, controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p < 0.0001, Regression, Linear; [statistical method as in outcome 5, analysis 4]; Slope = -30.23, 95% CI 2-sided [-43.23 to -17.23], Standard Error of Mean 6.25 — Effect of EMG-PR (compared to IMU group)

6. Secondary Outcome: Jebsen-Taylor Hand Function Test (JTHFT) 7 Subtests
Description: JTHFT Writing: Evaluates the time needed to print a 24-letter, third-grade reading difficulty sentence. JTHFT Page turning: Evaluates the time needed to turn over 7.6 x 12.7 cm (3x5") cards in simulated page turning. JTHFT Small objects: Evaluates the time needed to perform pick up small common objects including pennies, paper clips, bottle caps and placing them in a container. JTHFT Stacking checkers: Evaluates the time needed to stack four checkers. JTHFT Simulated feeding: Evaluates the time needed to perform simulated feeding. JTHFT Moving large empty cans: Evaluates the time needed to move large empty cans. JTHFT Moving large 1 lb. cans: Evaluates the time needed to move 1 lb. cans. All subtests are modified to cap the maximal time for the subtask at 120 seconds and is scored as the number of items completed per second.
Time Frame: as for outcome 2
Population: Prosthesis users only, at baseline, completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: items completed per second
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 33 | 11
items completed per second
  JTHFT Writing: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Writing: Prosthesis users at baseline | 0.37 (0.24) | 0.37 (0.17)
  JTHFT Writing: Completers at End of Part A | 0.35 (0.18) | 0.39 (0.12)
  JTHFT Writing: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Writing: Completers End of B | 0.45 (0.19) | 0.42 (0.16)
  JTHFT Page Turning: Prosthesis users at baseline: number analyzed (Participants) | 28 | 10
  JTHFT Page Turning: Prosthesis users at baseline | 0.09 (0.08) | 0.10 (0.03)
  JTHFT Page Turning: : Completers at End of Part A | 0.05 (0.04) | 0.06 (0.03)
  JTHFT Page Turning: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Page Turning: Completers End of B | 0.10 (0.07) | 0.07 (0.03)
  JTHFT Small Items: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Small Items: Prosthesis users at baseline | 0.08 (0.08) | 0.07 (0.06)
  JTHFT Lifting Small Items:: Completers End of Part | 0.07 (0.07) | 0.04 (0.03)
  JTHFT Lifting Small Items: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Lifting Small Items: Completers End of B | 0.08 (0.06) | 0.06 (0.06)
  JTHFT Checkers: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Checkers: Prosthesis users at baseline | 0.12 (0.08) | 0.12 (0.06)
  JTHFT Checkers: Completers End of Part A | 0.07 (0.06) | 0.06 (0.05)
  JTHFT Checkers: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Checkers: Completers End of B | 0.09 (0.08) | 0.11 (0.04)
  JTHFT Feeding: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Feeding: Prosthesis users at baseline | 0.11 (0.09) | 0.12 (0.06)
  JTHFT Feeding: Completers End of Part A | 0.07 (0.06) | 0.05 (0.05)
  JTHFT Feeding: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Feeding: Completers End of B | 0.10 (0.07) | 0.05 (0.03)
  JTHFT Light Cans: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Light Cans: Prosthesis users at baseline | 0.21 (0.15) | 0.22 (0.08)
  JTHFT Light Cans: Completers End of Part A | 0.19 (0.15) | 0.10 (0.08)
  JTHFT Light Cans: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Light Cans: Completers End of B | 0.24 (0.16) | 0.14 (0.06)
  JTHFT Heavy Cans: Prosthesis users at baseline: number analyzed (Participants) | 26 | 10
  JTHFT Heavy Cans: Prosthesis users at baseline | 0.24 (0.17) | 0.24 (0.11)
  JTHFT Heavy Cans: Completers End of Part A | 0.20 (0.15) | 0.13 (0.09)
  JTHFT Heavy Cans: Completers End of B: number analyzed (Participants) | 18 | 7
  JTHFT Heavy Cans: Completers End of B | 0.28 (0.15) | 0.16 (0.07)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Writing data at both time points); Test type: Superiority; p = 0.6691, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.05 to 0.07], Standard Deviation 0.17 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Page turning data at both time points); Test type: Superiority; p = 0.0511, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.05 to 0.00], Standard Deviation 0.06 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 3: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Lifting Small Items data at both time points); Test type: Superiority; p = 0.5942, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.02 to 0.04], Standard Deviation 0.09 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 4: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Checkers data at both time points); Test type: Superiority; p = 0.0101, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.07 to -0.01], Standard Deviation 0.08 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 5: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Feeding data at both time points); Test type: Superiority; p = 0.1063, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.06 to 0.01], Standard Deviation 0.09 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 6: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Light Cans data at both time points); Test type: Superiority; p = 0.2474, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.06 to 0.01], Standard Deviation 0.12 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 7: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with JTHFT: Heavy Cans data at both time points); Test type: Superiority; p = 0.1604, t-test, 2 sided; The sample for this paired t-test was 31 participants; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.09 to 0.02], Standard Deviation 0.14 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 8: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from JTHFT: Writing measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.4208, Regression, Linear; The sample for this analysis was 24 participants with TR or TH amputation level who completed data collection for JTHFT at End of Part B; Slope = -0.06, 95% CI 2-sided [-0.12 to 0.09], Standard Error of Mean 0.07 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 9: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from JTHFT: Page Turning measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.1959, Regression, Linear; The sample for this analysis was 23 participants with TR or TH amputation level who completed data collection for JTHFT at End of Part B; Slope = -0.04, 95% CI 2-sided [-0.09 to 0.02], Standard Error of Mean 0.03 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 10: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Test type: Superiority — Linear regression of scores from JTHFT: Lifting Small Items measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; p = 0.3328, Regression, Linear; [statistical method as in outcome 6, analysis 9]; Slope = -0.03, 95% CI 2-sided [-0.09 to 0.03], Standard Error of Mean 0.03 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 11: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from JTHFT: Checkers measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.6585, Regression, Linear; [statistical method as in outcome 6, analysis 9]; Slope = 0.01, 95% CI 2-sided [-0.05 to 0.08], Standard Error of Mean 0.03 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 12: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Test type: Superiority — Linear regression of scores from JTHFT: Feeding measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; p = 0.0552, Regression, Linear; [statistical method as in outcome 6, analysis 9]; Slope = -0.06, 95% CI 2-sided [-0.12 to 0.00], Standard Error of Mean 0.03 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 13: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from JTHFT: Light Cans measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0319, Regression, Linear; [statistical method as in outcome 6, analysis 9]; Slope = -0.13, 95% CI 2-sided [-0.25 to -0.01], Standard Error of Mean 0.06 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 14: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from JTHFT: Heavy Cans measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0073, Regression, Linear; [statistical method as in outcome 6, analysis 9]; Slope = -0.14, 95% CI 2-sided [-0.24 to -0.04], Standard Error of Mean 0.05 — Effect of EMG-PR (compared to IMU group)

7. Secondary Outcome: University of New Brunswick Test of Prosthetic Function (UNB)
Description: This test is performed with unilateral amputees only. The subtest used includes wrapping a parcel, sewing a button on cloth, cutting meat, drying dishes, sweeping floor, and using a dustpan and brush. Each task was rated for both spontaneity and skill. UNB Spontaneity: Spontaneity rates spontaneity of prosthesis use (0=prosthesis not used to 4=immediate, consistent use of terminal device. UNB Skill: rates skill of performing the activities (0 = prothesis not used to 4 = active terminal device is quick & smooth). Summary scores are calculated for each subscale by averaging items and range from 0 to 4 with higher scores reflecting higher spontaneity and skill.
Time Frame: as for outcome 2
Population: Prosthesis users only, at baseline, completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 31 | 11
score on a scale
  UNB Spontanaity: Prosthesis users at baseline: number analyzed (Participants) | 24 | 10
  UNB Spontanaity: Prosthesis users at baseline | 3.1 (0.5) | 3.2 (0.4)
  UNB Spontanaity: Completers End of Part A | 3.0 (0.4) | 3.1 (0.5)
  UNB Spontaneity: Completers End of Part B: number analyzed (Participants) | 16 | 7
  UNB Spontaneity: Completers End of Part B | 3.2 (0.4) | 3.4 (0.3)
  UNB Skill: Prosthesis users at baseline: number analyzed (Participants) | 24 | 10
  UNB Skill: Prosthesis users at baseline | 3.0 (0.5) | 3.0 (0.5)
  UNB Skill: Completers End of Part A | 2.8 (0.5) | 2.9 (0.5)
  UNB Skill: Completers End of Part B: number analyzed (Participants) | 16 | 7
  UNB Skill: Completers End of Part B | 3.1 (0.4) | 3.2 (0.3)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with UNB: Spontaneity data at both time points); Test type: Superiority; p = 0.6529, t-test, 2 sided; The sample for this paired t-test was 30 participants; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.24 to 0.15], Standard Deviation 0.52 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with UNB: Skill data at both time points); Test type: Superiority; p = 0.8490, t-test, 2 sided; The sample for this paired t-test was 30 participants; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.26 to 0.22], Standard Deviation 0.64 — Mean difference is the change in scores from baseline to End of A
Statistical Analysis 3: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from UNB: Spontaneity measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.4589, Regression, Linear; The sample for this analysis was 23 participants with TR or TH amputation level who completed data collection for UNB: Spontaneity at End of Part B; Slope = 0.13, 95% CI 2-sided [-0.22 to 0.48], Standard Error of Mean 0.17 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 4: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from UNB: Skill measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.7110, Regression, Linear; The sample for this analysis was 23 participants with TR or TH amputation level who completed data collection for UNB: Skill at End of Part B; Slope = 0.07, 95% CI 2-sided [-0.31 to 0.44], Standard Error of Mean 0.18 — Effect of EMG-PR (compared to IMU group)

8. Secondary Outcome: Timed Measure of Activity Performance (T-MAP)
Description: The T-MAP is a performance measure of daily activities for persons with upper limb amputation utilizing 5 every day activities. Time (seconds) to completion of activity is measured and summed to obtain overall timed score. Lower overall scores (less time taken) indicate better / faster activity performance
Time Frame: as for outcome 2
Population: Baseline participants and completers at End of A and End of B
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 39 | 13
Seconds
  Prosthesis users at baseline | 459.8 (223.6) | 366.5 (108.5)
  Completers End of Part A: number analyzed (Participants) | 29 | 9
  Completers End of Part A | 748.1 (461.7) | 549.0 (257.5)
  Completers End of Part B: number analyzed (Participants) | 14 | 6
  Completers End of Part B | 624.8 (429.1) | 443.3 (154.2)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data for participants at baseline and completers at End of A (i.e participants with T-MAP data at both time points); Test type: Superiority; p < 0.0001, t-test, 2 sided; The sample for this paired t-test was 38 participants; Mean Difference (Net) = 253.6, 95% CI 2-sided [146.7 to 360.5], Standard Deviation 325.2; Mean difference is the change in scores from Baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from T-MAP measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.3397, Regression, Linear; The sample for this analysis was 22 participants with TR or TH amputation level who completed data collection for T-MAP at End of Part B; Slope = -183.1, 95% CI 2-sided [-574.3 to 208.2], Standard Error of Mean 186.9 — Effect of EMG-PR (compared to IMU group)

9. Secondary Outcome: Upper Extremity Functional Scale (UEFS) From the Orthotics and Prosthetics Users Survey (OPUS)
Description: The UEFS is a self-report measure developed for use with upper limb adult amputees. It includes 23 activities: selfcare, instrumental, and daily living tasks using a 5-point scale from 1=Very Easy to 5=Cannot perform. Total score was calculated using IRT methods and ranged from 0 to 100 with lower scores reflecting better function.
Time Frame: as for outcome 2
Population: Baseline participants and completers at End of A and End of B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 27 | 10
score on a scale
  Prosthesis users at baseline: number analyzed (Participants) | 22 | 10
  Prosthesis users at baseline | 42.4 (8.1) | 37.6 (14.9)
  Completers End of Part A: number analyzed (Participants) | 27 | 9
  Completers End of Part A | 44.3 (6.3) | 45.8 (8.2)
  Completers End of Part B: number analyzed (Participants) | 14 | 5
  Completers End of Part B | 38.0 (9.5) | 41.5 (8.3)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0465, t-test, 2 sided; The sample for this paired t-test was 24 participants; Mean Difference (Net) = 4.30, 95% CI 2-sided [0.07 to 8.53], Standard Deviation 10.01 — Mean difference is the change in scores from Baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from UEFS measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.3450, Regression, Linear; The sample for this analysis was 19participants with TR or TH amputation level who completed data collection for UEFS at End of Part B; Slope = -2.39, 95% CI 2-sided [-7.60 to 2.82], Standard Error of Mean 2.46 — Effect of EMG-PR (compared to IMU group)

10. Secondary Outcome: The Community Reintegration of Service Members Computer Adaptive Test (CRIS-CAT)
Description: The CRIS measures community reintegration. It consists of three scales extent and frequency, perceived limitations, and satisfaction. Higher scores (range 0-100) indicate better community integration.
Time Frame: as for outcome 2
Population: Baseline participants and completers at End of A and End of B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
Number analyzed (Participants) | 38 | 13
score on a scale
  CRIS Extent of Participation: Baseline | 53.8 (8.1) | 53.1 (9.1)
  CRIS Extent: Completers End of Part A: number analyzed (Participants) | 33 | 11
  CRIS Extent: Completers End of Part A | 54.4 (10.3) | 52.4 (8.2)
  CRIS Extent: Completers End of Part B: number analyzed (Participants) | 19 | 7
  CRIS Extent: Completers End of Part B | 58.1 (9.4) | 51.3 (8.6)
  CRIS Perceived Limitations: Baseline | 53.7 (12.9) | 49.8 (6.6)
  CRIS Perceived: Completers End of Part A: number analyzed (Participants) | 33 | 11
  CRIS Perceived: Completers End of Part A | 53.5 (12.5) | 49.5 (5.8)
  CRIS Perceived: Completers End of Part B: number analyzed (Participants) | 19 | 7
  CRIS Perceived: Completers End of Part B | 59.5 (17.1) | 47.6 (4.6)
  CRIS Satisfaction: Baseline | 54.0 (11.2) | 48.6 (6.5)
  CRIS Satisfaction: Completers End of Part A: number analyzed (Participants) | 33 | 11
  CRIS Satisfaction: Completers End of Part A | 52.0 (7.7) | 48.3 (4.7)
  CRIS Satisfaction: Completers End of Part B: number analyzed (Participants) | 19 | 7
  CRIS Satisfaction: Completers End of Part B | 55.1 (12.7) | 48.7 (5.7)
Statistical Analysis 1: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data for participants at baseline and completers at End of A (i.e participants with CRIS: Extent of Limitations data at both time points); Test type: Superiority; p = 0.6881, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = 0.47, 95% CI 2-sided [-1.86 to 2.79], Standard Deviation 7.54 — Mean difference is the change in scores from Baseline to End of A
Statistical Analysis 2: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with CRIS: Perceived Limitations data at both time points); Test type: Superiority; p = 0.7363, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -0.72, 95% CI 2-sided [-5.01 to 3.67], Standard Deviation 13.95 — Mean difference is the change in scores from Baseline to End of A
Statistical Analysis 3: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Pairwise t-test for data from prosthesis users at baseline and completers at End of A (i.e. participants with CRIS: Satisfaction data at both time points); Test type: Superiority; p = 0.2361, t-test, 2 sided; The sample for this paired t-test was 43 participants; Mean Difference (Net) = -1.49, 95% CI 2-sided [-3.99 to 1.01], Standard Deviation 8.12 — Mean difference is the change in scores from Baseline to End of A
Statistical Analysis 4: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from CRIS-CAT: Extent of Limitations measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0932, Regression, Linear; The sample for this analysis was 24 participants with TR or TH amputation level who completed data collection for CRIS-CAT at End of Part B; Slope = -7.07, 95% CI 2-sided [-15.43 to 1.29], Standard Error of Mean 4.02 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 5: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from CRIS-CAT: Perceived Limitations measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.0951, Regression, Linear; [statistical method as in outcome 10, analysis 4]; Mean Difference (Final Values) = -10.5, 95% CI 2-sided [-22.9 to 1.99], Standard Error of Mean 6.0 — Effect of EMG-PR (compared to IMU group)
Statistical Analysis 6: Comparison: Advanced Upper Limb Prosthetic Device IMU Controlled vs Advanced Upper Limb Prosthetic EMG-PR Controlled; Linear regression of scores from CRIS-CAT: Satisfaction measure at 9-12 weeks (End of B), comparing groups by control type, and controlling for amputation level (transhumeral or transradial). Persons with shoulder level devices are excluded from this analysis; Test type: Superiority; p = 0.2346, Regression, Linear; [statistical method as in outcome 10, analysis 4]; Slope = -4.91, 95% CI 2-sided [-13.3 to 3.43], Standard Error of Mean 4.01 — Effect of EMG-PR (compared to IMU group)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected non-systematically as events were reported. They were also summarized at annual IRB continuing reviews from baseline to after 9-12 weeks of home use.
Description: Definitions of adverse events are consistent with clinicaltrials.gov definitions.
Arm/Group | Advanced Upper Limb Prosthetic Device IMU Controlled | Advanced Upper Limb Prosthetic EMG-PR Controlled
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/13
Other Adverse Events (participants affected / at risk) | 5/39 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Upper Limb Prosthetic Device IMU Controlled (N=39) | Advanced Upper Limb Prosthetic EMG-PR Controlled (N=13)
Unrelated adverse event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject hospitalized due to an unrelated cellulitis flare-up in his lower limb
Unrelated adverse event (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject was in a car accident in a rental car on his way to the airport after the study had ended
Adverse Event (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject had a skin irritation, possibly due to socket wear
Adverse event (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Musculoskeletal pain related to wearing or using the device: including back or ankle pain
Adverse event (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject was using the prosthesis to eat with a fork and sustained a minor cut to his lip.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT01551420/Prot_SAP_000.pdf